CLINICAL TRIAL: NCT03987763
Title: A Phase 4, Open-Label, Multicenter Study Evaluating the Absorption and Systemic Pharmacokinetics and HPA Axis Suppression Potential of Topically Applied IDP-122 Lotion in Pediatric Subjects With Moderate to Severe Plaque Psoriasis
Brief Title: A Safety and Pharmacokinetics Study of IDP-122 Lotion in Pediatric Participants With Plaque Psoriasis
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: V01-122A-401
Record Dates: First submitted 2019-06-13; First posted 2019-06-17 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Psoriasis
Keywords: Plaque psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- IDP-122 Lotion (Experimental): Two cohorts of pediatric participants (1 cohort of participants age 12 to 16 years 11 months and 1 cohort of participants age 6 to 11 years 11 months) will apply IDP-122 Lotion to Investigator identified lesions affecting a minimum of 10% body surface area (BSA) once daily for 8 weeks.
  Interventions: Drug: IDP-122 Lotion

INTERVENTIONS:
Drug: IDP-122 Lotion — Topical

SUMMARY:
This study is to evaluate the safety, the systemic exposure of halobetasol propionate (HP), and the hypothalamic-pituitary-adrenal (HPA) axis suppression potential for topically applied IDP-122 lotion in pediatric participants with moderate to severe plaque psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Is 6 to 16 years 11 months of age at time of informed consent/assent obtained.
* Verbal and written informed consent/assent obtained from the participant and/or parent or legal guardian.
* Has a clinical diagnosis of psoriasis at Screening and Baseline with an Investigator's Global Assessment (IGA) score of 3 or 4. The face, scalp, axillae, and intertriginous areas are to be excluded in this assessment, if psoriasis is present.
* Has an area of plaque psoriasis appropriate for topical treatment that involves a BSA of at least 10% at Screening and Baseline. The face, scalp, axillae, and intertriginous areas are to be excluded in this calculation.
* Is willing and able to avoid prolonged exposure of the treatment area to ultraviolet radiation (natural and artificial) for the duration of the study.
* Is in good general adrenal health, as determined by a 30-minute postcosyntropin stimulation serum cortisol level that is >18 μg/dL at the Screening visit.
* Females of childbearing potential and females who are pre-menses (9 years and older) must be willing to practice effective contraception for the duration of the study.

Exclusion Criteria:

* Has a history of adrenal disease.
* Presents with any concurrent skin condition that could interfere with the evaluation of the treatment areas, as determined by the Investigator.
* Is pregnant, nursing an infant, or planning a pregnancy during the study period.
* Has received treatment with any investigational drug or device within 60 days or 5 drug half-lives (whichever is longer) prior to baseline or is concurrently participating in another clinical study with an investigational drug or device.
* Received treatment with a topical antipsoriatic drug product other than corticosteroids within 14 days prior to the Baseline visit and/or treatment containing corticosteroids within 28 days prior to the screening HPA axis stimulation test.
* Has a history of hypersensitivity or allergic reaction to any of the study drug constituents.
* Is considered by the Investigator, for any other reason, to be an unsuitable candidate for the study.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Estimated)
Dates: Start 2019-10-22 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics: Maximum Observed Drug (Halobetasol Propionate) Concentration in Plasma (Cmax) of IDP-122 Lotion Analytes | 0 (predose), 1, 2, 4, 8, 12, and 24 hours postdose
  On Days 28-29, blood samples will be collected from each participant for the determination of plasma concentrations and PK parameters of IDP-122 Lotion analytes.

SECONDARY OUTCOMES:
Proportion of Participants With Hypothalamic-Pituitary-Adrenal (HPA) Axis Suppression | Week 8
  An HPA axis suppression is defined as a 30 minute poststimulation cortisol level of ≤18 micrograms/deciliter (μg/dL) at the end of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Alison Magnotti-Nagel, Study Director — Bausch Health
Locations (9):
- United States (7):
  - Bausch Site 11, Fountain Valley, California
  - Bausch Site 2, Thousand Oaks, California
  - Bausch Site 07, Doral, Florida
  - Bausch Site 3, Miami, Florida
  - Bausch Site 06, Miami, Florida
  - Bausch Site 05, Spartanburg, South Carolina
  - Bausch Site 1, Spokane, Washington
- Bausch Site 12, Santo Domingo, Dominican Republic
- Bausch Site 4, Panama City, Panama